CLINICAL TRIAL: NCT01383304
Title: Is a Reduced Biochemical Response to Aspirin Associated With Increased Cardiovascular Morbidity and Mortality in High Risk Patients With Coronary Artery Disease?
Brief Title: Aspirin Response in High Risk Patients With Coronary Artery Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital Skejby (Other); Danish Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 22527
Record Dates: First submitted 2011-06-22; First posted 2011-06-28 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Coronary Artery Disease; Myocardial Infarction; Diabetes Mellitus; Renal Insufficiency, Chronic
Keywords: Platelet aggregation; Aspirin; Drug resistance; Thromboxane B2; Pharmacologic Actions; Platelet Aggregation Inhibitors
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Diabetes Mellitus; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma, urine
Oversight: Data Monitoring Committee: No

SUMMARY:
Previous studies indicate that patients with cardiovascular disease have a variable response to aspirin. Despite treatment with aspirin a large number of patients suffer a myocardial infarction. This has given rise to the phenomenon "aspirin low-responsiveness". Laboratory aspirin low-responsiveness can be defined as the failure of aspirin to inhibit platelet production of thromboxane A2 or inhibit thromboxane-dependent platelet aggregation. Whether a low platelet response to aspirin results in an increased risk of future thrombotic events is of great clinical significance, but is still unknown.

The investigators hypothesize that patients with a reduced response to aspirin, determined by platelet aggregation using the apparatus Verify Now Aspirin and Multiplate, have a higher risk of thrombosis.

The purpose of this study is to investigate whether a higher incidence of cardiovascular events is found in patients with coronary artery disease (CAD) having a reduced biochemical response to aspirin compared with CAD patients having a normal biochemical response to aspirin. In addition to CAD, all patients have at least one of the following risc factors: previous myocardial infarction, type 2 diabetes mellitus and/or renal insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease verified by coronary angiogram
* Treatment with aspirin 75 mg/d for at least the previous 7 days
* Previous myocardial infarction more than one year ago (groups with previous myocardial infarction)
* Type 2 diabetes mellitus treated with oral antidiabetics and/or insulin (groups with type 2 diabetes mellitus)
* Renal insufficiency; glomerular filtration rate <60 ml/min at the time of blood sampling (groups with renal insufficiency)

Exclusion Criteria:

* Treatment with NSAIDs, clopidogrel, ticlopidine, dipyridamole, warfarin or any other drugs known to affect platelet function
* Ischemic vascular event within the previous 12 months
* Revascularization (angioplasty or coronary by-pass graft surgery) within the previous 12 months
* Platelet count <120 x 10^9/L or >450 x 10^9/L
* For patients without diabetes: fast glucose >7 mmol/L
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 906 patients with CAD. In addition to CAD, all patients have at least one of the following risc factors: previous myocardial infarction, type 2 diabetes mellitus and/or renal insufficiency.
  Eligible patients are identified in the Western Denmark Heart Registry.
Sampling Method: Non-Probability Sample
Enrollment: 906 (Actual)
Dates: Start 2007-11; Primary Completion 2011-01 (Actual); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Combined primary endpoint: Cardiovascular death, acute myocardial infarction, ischaemic stroke | Evaluation after 3 years

SECONDARY OUTCOMES:
Combined secondary endpoint: Cardiovascular death, acute myocardial infarction, ischaemic stroke | Evaluation after 5 years
Single endpoints:cardiovascular death; acute myocardial infarction; ischemic stroke; stent thrombosis; all-cause death | Evaluation after 3 and 5 years

OTHER OUTCOMES:
Genotype according to pre-specified genetic single nucleotide polymorphisms (SNPs) | Baseline
  At the day of blood sampling, plasma samples are retrieved for DNA extraction. DNA samples are used to evaluate if pre-specified genetic single nucleotide polymorphisms (SNPs) are associated with platelet aggregation levels.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Mette Hvas, MD, Ph.D, Principal Investigator — Department of Clinical Biochemistry, Aarhus University Hospital, Skejby, Denmark
Locations (1):
- Department of Clinical Biochemistry, Aarhus University Hospital, Skejby, Aarhus N, Denmark

REFERENCES:
- [Background] Nielsen HL, Kristensen SD, Thygesen SS, Mortensen J, Pedersen SB, Grove EL, Hvas AM. Aspirin response evaluated by the VerifyNow Aspirin System and light transmission aggregometry. Thromb Res. 2008;123(2):267-73. doi: 10.1016/j.thromres.2008.03.023. Epub 2008 May 21. PMID 18499236
- [Background] Pedersen SB, Grove EL, Nielsen HL, Mortensen J, Kristensen SD, Hvas AM. Evaluation of aspirin response by Multiplate whole blood aggregometry and light transmission aggregometry. Platelets. 2009 Sep;20(6):415-20. doi: 10.1080/09537100903100643. PMID 19658002
- [Background] Hedegaard SS, Hvas AM, Grove EL, Refsgaard J, Rocca B, Davi G, Kristensen SD. Optical platelet aggregation versus thromboxane metabolites in healthy individuals and patients with stable coronary artery disease after low-dose aspirin administration. Thromb Res. 2009 May;124(1):96-100. doi: 10.1016/j.thromres.2008.12.034. Epub 2009 Feb 11. PMID 19215971
- [Background] Grove EL, Hvas AM, Johnsen HL, Hedegaard SS, Pedersen SB, Mortensen J, Kristensen SD. A comparison of platelet function tests and thromboxane metabolites to evaluate aspirin response in healthy individuals and patients with coronary artery disease. Thromb Haemost. 2010 Jun;103(6):1245-53. doi: 10.1160/TH09-08-0527. Epub 2010 Mar 29. PMID 20352155
- [Background] Mortensen SB, Larsen SB, Grove EL, Kristensen SD, Hvas AM. Reduced platelet response to aspirin in patients with coronary artery disease and type 2 diabetes mellitus. Thromb Res. 2010 Oct;126(4):e318-22. doi: 10.1016/j.thromres.2010.03.013. Epub 2010 May 7. PMID 20451957
- [Result] Larsen SB, Neergaard-Petersen S, Grove EL, Kristensen SD, Hvas AM. Increased platelet aggregation and serum thromboxane levels in aspirin-treated patients with prior myocardial infarction. Thromb Haemost. 2012 Jul;108(1):140-7. doi: 10.1160/TH12-01-0026. Epub 2012 Apr 26. PMID 22534977
- [Derived] Wurtz M, Nissen PH, Grove EL, Kristensen SD, Hvas AM. Genetic determinants of on-aspirin platelet reactivity: focus on the influence of PEAR1. PLoS One. 2014 Oct 31;9(10):e111816. doi: 10.1371/journal.pone.0111816. eCollection 2014. PMID 25360888